CLINICAL TRIAL: NCT00045591
Title: Evaluation Of Novel Therapeutic Agents (Celecoxib: NSC # 719627) Against Breast Cancer: An Innovative Randomized Phase II Trial Design
Brief Title: Celecoxib in Treating Women With Metastatic or Recurrent Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CALGB-40105; U10CA031946 (NIH); CALGB-40105; CDR0000256905 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib 100 mg (Experimental)
  Interventions: Drug: celecoxib
- Celecoxib 400 mg (Experimental)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: celecoxib — 100 mg PO bid
  Arms: Celecoxib 100 mg
Drug: Celecoxib — 400 mg PO bid
  Arms: Celecoxib 400 mg

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for their growth and by stopping blood flow to the tumor. It is not yet known which regimen of celecoxib is more effective in treating breast cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of two regimens of celecoxib in treating women who have metastatic or recurrent breast cancer

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival of women with metastatic or recurrent breast cancer treated with 2 dose levels of celecoxib.

Secondary

* Compare the side effects of the 2 dose levels of this drug in these patients.
* Compare the overall survival of patients treated with the 2 dose levels of this drug.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to disease status at study entry (complete response vs partial response vs stable) and prior metastatic/recurrent chemotherapy regimens (1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral high-dose celecoxib twice daily.
* Arm II: Patients receive oral low-dose celecoxib twice daily. In both arms, treatment continues until first disease progression. At disease progression, treatment assignment is unblinded and treatment may continue at the treating physician's discretion. Patients initially randomized to the low-dose arm may either continue on that dosage or crossover to the high-dose arm. Patients initially randomized to the high-dose arm may continue on that dosage. Treatment after disease progression may continue for up to 12 months.

Patients are followed every 3 months for 1 year and then every 6 months for up to 4 years.

PROJECTED ACCRUAL: A total of 132 patients (88 in the high-dose arm and 44 in the low-dose arm) will be accrued for this study within 22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Metastatic or recurrent disease documented by physical or radiographic examination
  * Isolated recurrence of breast cancer not considered eligible
  * Bone disease alone allowed
* At least 4 prior courses (or 4 months) of chemotherapy resulting in stable disease, partial response, or complete response
* Treated brain metastases allowed provided all of the following conditions are met:

  * Palliation achieved without evidence of progression for at least 3 months after completion of radiotherapy and/or surgical treatment
  * At least 30 days since prior dexamethasone or other corticosteroids
  * Documentation of another site of metastatic disease (in addition to brain metastases)
* Measurable or evaluable disease
* Pleural or peritoneal effusion as only manifestation of disease allowed if palliated by prior chemotherapy
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* CTC (ECOG) 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 2.5 times ULN (5 times ULN if liver metastases present)
* Albumin at least 3.0 g/dL

Renal

* Creatinine no greater than 1.5 times ULN

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other active malignancy within the past 2 years except nonmelanoma skin cancer
* No active peptic ulcer disease
* No known hypersensitivity to sulfonamides, aspirin, or other NSAIDs, including celecoxib

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Concurrent trastuzumab (Herceptin) allowed if initiated at least 3 months prior to study entry

Chemotherapy

* See Disease Characteristics
* At least 6 weeks since prior chemotherapy
* No more than 2 prior chemotherapy regimens for recurrent or metastatic disease

Endocrine therapy

* See Disease Characteristics
* Prior hormonal therapy for metastatic disease allowed
* No concurrent hormonal therapy except hormones for noncancer-related conditions (e.g., insulin for diabetes)

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* Prior radiotherapy to the breast and for metastatic disease allowed
* No concurrent palliative radiotherapy

Surgery

* See Disease Characteristics

Other

* Prior adjuvant therapy for metastatic disease allowed
* Concurrent bisphosphonates allowed
* Concurrent low-dose aspirin (no greater than 325 mg/day) is allowed
* No other concurrent therapy with celecoxib or other nonsteroidal anti-inflammatory drugs (NSAIDs) (e.g., rofecoxib, aspirin, choline magnesium trisalicylate, ibuprofen, naproxen, etodolac, oxaprozin, diflunisal, nabumetone, or tolmetin)
* No concurrent fluconazole

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-02; Primary Completion 2005-08 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Shapiro, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (74):
- United States (74):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Lagrange Oncology Associates, La Grange, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Comprehensive Cancer Center at Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia